CLINICAL TRIAL: NCT06102018
Title: Diagnostic Biomarkers Exploration of Breast Cancer From Serum and Urine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-149-02
Record Dates: First submitted 2023-05-09; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasm Female
Keywords: Serum and Urine Biomarkers,Machine Learning,Diagnostic Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood sample contains DNA, but the measurement does not involve DNA. Once the project is complete, the sample will be properly disposed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast cancer patients: No intervention. The patients who are diagnosed as breast cancer by postoperative pathological.
  Interventions: Diagnostic Test: Collect blood and urine，pathological specimens if necessary
- Patients with benign breast lesions: No intervention. The patients who are diagnosed asbenign breast lesions by postoperative pathological.
  Interventions: Diagnostic Test: Collect blood and urine，pathological specimens if necessary
- Healthy population: No intervention. The volunteers.
  Interventions: Diagnostic Test: Collect blood and urine，pathological specimens if necessary

INTERVENTIONS:
Diagnostic Test: Collect blood and urine，pathological specimens if necessary — Use EDTA anticoagulant pipe to collect all blood 2ml, and collect 3ml of urine with sterile test tube

SUMMARY:
The goal of this observational study is to find the diagnostic biomarkers in serum and urine from early breast cancer patients. The main questions it aims to answer are:

* compare the different biomarkers in serum and urine from breast cancer patients, benign lesions and healthy population.
* construct the best diagnostic model by machine learning to distinguish breast cancer and non-breast cancer patients.

Participants, including breast and non-breast cancer patients will be asked to provides blood and urine during their diagnosis and treatment process without changing the original treatment. When necessary, specimens will be collected during the surgery，without affecting pathological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Signing the consent of informedness;
2. Patients with breast mass who need surgery after examination;
3. Cardiac ultrasound indicates that the blood score of the heart is within the normal range;
4. ECOG≤0-2 points;
5. Oversure function is acceptable.

Exclusion Criteria:

1. Merge other malignant tumors such as gynecologic oncology;
2. After evaluation, the internal organs are not suitable.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: early breast cancer(Tis,T1-3N0-1M0)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The different biomarkers in malignant and benign breast diseases | It is expected to be one to two years.
  By analyzing the differences (eg:PCA, FC and et al.)in the composition of proteins in blood and urine, biomarkers with significant differences between the two groups will be obtained.
Diagnostic models used different biomarkers by machine learning | Within half a year after the completion of the test.
  Using biomarkers that detect discrepancies, combined with machine learning to build early breast cancer diagnostic models.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China